CLINICAL TRIAL: NCT01484496
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, 52-Week Study to Evaluate the Efficacy and Safety of Belimumab (HGS1006) Administered Subcutaneously (SC) to Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: A Study of Belimumab Administered Subcutaneously in Subjects With Systemic Lupus Erythematosus (SLE)
Acronym: BLISS-SC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Human Genome Sciences Inc., a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112341; 2011-003814-18; HGS1006-C1115
Record Dates: First submitted 2011-11-28; First posted 2011-12-02 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Subcutaneous; Lupus; Systemic Lupus Erythematosus; SLE; Belimumab; Autoimmune Disease; Antibodies
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases | interventions — belimumab; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo plus standard therapy (Placebo Comparator): Placebo SC plus standard therapy; placebo administered on Day 0 and then weekly (ie, every 7 days) through Week 51, with final evaluation at Week 52 in the double-blind period. In the open-label extension period, placebo subjects who opt to participate will receive belimumab 200 mg SC weekly for an additional 6-months.
  Interventions: Biological: Placebo; Drug: Standard therapy
- Belimumab 200 mg SC plus standard therapy (Experimental): Belimumab 200 mg SC plus standard therapy; belimumab administered on Day 0 and then weekly (ie, every 7 days) through Week 51, with a final evaluation at Week 52 in the double-blind period. In the open-label extension period, subjects who opt to participate will continue on the same dose of belimumab for an additional 6-months.
  Interventions: Biological: Belimumab 200 mg SC; Drug: Standard therapy

INTERVENTIONS:
Biological: Placebo — Placebo
  Arms: Placebo plus standard therapy
Biological: Belimumab 200 mg SC — Belimumab 200 mg SC
  Other Names: BENLYSTA™
  Arms: Belimumab 200 mg SC plus standard therapy
Drug: Standard therapy — Standard therapy comprises any of the following (alone or in combination): corticosteroids, antimalarials, non-steroidal anti-inflammatory drugs (NSAIDs), and immunosuppressives; biologics and intravenous cyclophosphamide are not permitted.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of belimumab administered subcutaneously (SC) to adult subjects with Systemic Lupus Erythematosus (SLE).

DETAILED DESCRIPTION:
This is a Phase 3, multi-center, international, randomized, double-blind, placebo-controlled, 52-week study to evaluate the efficacy, safety and tolerability of belimumab administered subcutaneously (SC) (200 mg weekly) in adult subjects with active Systemic Lupus Erythematosus (SLE). Approximately 816 SLE subjects will be randomized, with a target of about 544 subjects receiving belimumab and 272 subjects receiving placebo. Subjects completing the 52-week double-blind period can enter a 6-month open-label extension in which all subjects receive belimumab 200 mg SC weekly.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Clinical diagnosis of Systemic Lupus Erythematosus (SLE) by ACR criteria.
3. Active SLE disease.
4. Autoantibody-positive.
5. On stable SLE treatment regimen which may include corticosteroids (for example, prednisone), antimalarial (for example, hydroxychloroquine) and/or immunosuppressants (for example, azathioprine, methotrexate, mycophenolate, etc.)

Exclusion Criteria:

1. Pregnant or nursing.
2. Have received treatment with any B cell targeted therapy (for example, rituximab or belimumab).
3. Have received treatment an investigational biological agent in the past year.
4. Have received intravenous (IV) cyclophosphamide within 90 days of Day 0.
5. Have severe active lupus kidney disease.
6. Have severe active central nervous system (CNS) lupus.
7. Have required management of acute or chronic infections within the past 60 days.
8. Have current drug or alcohol abuse or dependence.
9. Have a positive test for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
10. Have a history of hypersensitivity reactions to contrast agents or biological medicines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 839 (Actual)
Dates: Start 2011-11-16; Primary Completion 2015-02-13 (Actual); Study Completion 2015-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (176):
- United States (71):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Peoria, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, San Leandro, California
  - GSK Investigational Site, Tustin, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Bridgeport, Connecticut
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Duluth, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Cumberland, Maryland
  - GSK Investigational Site, Hagerstown, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Saint Clair Shores, Michigan
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Cruces, New Mexico
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Lake Success, New York
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Smithtown, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Bethlehem, Pennsylvania
  - GSK Investigational Site, Duncansville, Pennsylvania
  - GSK Investigational Site, Wyomissing, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Jackson, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Nassau Bay, Texas
  - GSK Investigational Site, Royalty, Texas
  - GSK Investigational Site, Arlington, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
  - GSK Investigational Site, Pennsylvania, Wyoming
- Argentina (3):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma Buenos Aires
- GSK Investigational Site, Vienna, Austria
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Liège
- Brazil (7):
  - GSK Investigational Site, Cuiabá, Mato Grosso
  - GSK Investigational Site, Juiz de Fora, Minas Gerais
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, Salvador
  - GSK Investigational Site, São Paulo
- Bulgaria (3):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
- Chile (3):
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Viña del Mar
- Colombia (4):
  - GSK Investigational Site, Barranquilla
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Bucaramanga
  - GSK Investigational Site, Medellín
- Croatia (3):
  - GSK Investigational Site, Osijek
  - GSK Investigational Site, Rijeka
  - GSK Investigational Site, Zagreb
- Czechia (2):
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Zlín
- Denmark (2):
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Odense C
- France (5):
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Suresnes
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- Germany (7):
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Bad Nauheim, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Hamburg
- Hungary (2):
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Zalaegerszeg
- Italy (3):
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Padua, Veneto
  - GSK Investigational Site, Genova
- Japan (7):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- Malaysia (2):
  - GSK Investigational Site, Kuala Lumpur
  - GSK Investigational Site, Seremban, Negeri Sembilan
- Mexico (5):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Cuernavaca, Morelos
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, México
  - GSK Investigational Site, San Luis Potosí City
- Philippines (6):
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Davao City
  - GSK Investigational Site, Iloilo City
  - GSK Investigational Site, Las Piñas
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Quezon City
- Poland (4):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Wroclaw
- Portugal (5):
  - GSK Investigational Site, Almada
  - GSK Investigational Site, Amadora
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
- GSK Investigational Site, Bucharest, Romania
- Russia (3):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Yaroslavl
- GSK Investigational Site, Belgrade, Serbia
- GSK Investigational Site, Singapore, Singapore
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Granada
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Stockholm
- Taiwan (4):
  - GSK Investigational Site, Gueishan Township,Taoyuan County
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
- Thailand (5):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Rajathevee
  - GSK Investigational Site, Ratchatewi
  - GSK Investigational Site, Songkhla
- Ukraine (6):
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Poltava
  - GSK Investigational Site, Vinnytsia
  - GSK Investigational Site, Zaporizhzhia
- United Kingdom (3):
  - GSK Investigational Site, Coventry, Warwickshire
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Nikolopoulos D, Cetrez N, Lindblom J, Parodis I. Neuropsychiatric involvement in systemic lupus erythematosus contributes to organ damage beyond the nervous system: a post-hoc analysis of 5 phase III randomized clinical trials. Rheumatol Int. 2024 Sep;44(9):1679-1689. doi: 10.1007/s00296-024-05667-5. Epub 2024 Aug 8. PMID 39115551
- [Derived] Jagerback S, Gomez A, Parodis I. Predictors of renal flares in systemic lupus erythematosus: a post-hoc analysis of four phase III clinical trials of belimumab. Rheumatology (Oxford). 2025 Feb 1;64(2):623-631. doi: 10.1093/rheumatology/keae023. PMID 38216728
- [Derived] Gomez A, Jagerback S, Sjowall C, Parodis I. Belimumab and antimalarials combined against renal flares in patients treated for extra-renal systemic lupus erythematosus: results from 4 phase III clinical trials. Rheumatology (Oxford). 2024 Feb 1;63(2):338-348. doi: 10.1093/rheumatology/kead253. PMID 37228028
- [Derived] Brunner HI, Abud-Mendoza C, Mori M, Pilkington CA, Syed R, Takei S, Viola DO, Furie RA, Navarra S, Zhang F, Bass DL, Eriksson G, Hammer AE, Ji BN, Okily M, Roth DA, Quasny H, Ruperto N. Efficacy and safety of belimumab in paediatric and adult patients with systemic lupus erythematosus: an across-study comparison. RMD Open. 2021 Sep;7(3):e001747. doi: 10.1136/rmdopen-2021-001747. PMID 34531304
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Maslen T, Bruce IN, D'Cruz D, Ianosev M, Bass DL, Wilkinson C, Roth DA. Efficacy of belimumab in two serologically distinct high disease activity subgroups of patients with systemic lupus erythematosus: post-hoc analysis of data from the phase III programme. Lupus Sci Med. 2021 Feb;8(1):e000459. doi: 10.1136/lupus-2020-000459. PMID 33568389
- [Derived] Lokhandwala T, Yue B, Coutinho AD, Bell CF. Within-trial economic analysis of flare data from the BLISS-SC trial of subcutaneous belimumab in systemic lupus erythematosus. Lupus Sci Med. 2021 Feb;8(1):e000438. doi: 10.1136/lupus-2020-000438. PMID 33558436
- [Derived] Doria A, Bass D, Schwarting A, Hammer A, Gordon D, Scheinberg M, Fox NL, Groark J, Stohl W, Kleoudis C, Roth D. A 6-month open-label extension study of the safety and efficacy of subcutaneous belimumab in patients with systemic lupus erythematosus. Lupus. 2018 Aug;27(9):1489-1498. doi: 10.1177/0961203318777634. Epub 2018 May 28. PMID 29807477
- [Derived] Doria A, Stohl W, Schwarting A, Okada M, Scheinberg M, van Vollenhoven R, Hammer AE, Groark J, Bass D, Fox NL, Roth D, Gordon D. Efficacy and Safety of Subcutaneous Belimumab in Anti-Double-Stranded DNA-Positive, Hypocomplementemic Patients With Systemic Lupus Erythematosus. Arthritis Rheumatol. 2018 Aug;70(8):1256-1264. doi: 10.1002/art.40511. Epub 2018 Jun 15. PMID 29671280
- [Derived] Stohl W, Schwarting A, Okada M, Scheinberg M, Doria A, Hammer AE, Kleoudis C, Groark J, Bass D, Fox NL, Roth D, Gordon D. Efficacy and Safety of Subcutaneous Belimumab in Systemic Lupus Erythematosus: A Fifty-Two-Week Randomized, Double-Blind, Placebo-Controlled Study. Arthritis Rheumatol. 2017 May;69(5):1016-1027. doi: 10.1002/art.40049. Epub 2017 Apr 7. PMID 28118533
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 112341 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112341 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112341 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112341 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112341 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112341 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112341 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (Par.) with active systemic lupus erythematosus (SLE) and who were on appropriate stable standard SLE therapy for a period of at least 30 days prior to Day 0 before entering the study were eligible for participation in the study.
Pre-assignment Details: A total of 1427 par. were screened, out of these 588 par. were screen failures and 839 par. were randomized, of which 836 par. received at least one dose of study treatment. Par. who successfully completed the initial 52-week Double-blind Phase had a choice to enter into a 6-month Open-label Extension Phase of this study.
Groups:
- Placebo SC: Par. received placebo administered subcutaneously (SC) once weekly through 51 weeks of thetreatment period. Par. continued with the stable standard therapy they were receiving during the Screening Period.
- Belimumab 200 mg SC: Par. received belimumab 200 milligrams (mg) administered SC once weekly through 51 weeks of the treatment period. Par. continued with the stable standard therapy they were receiving during the Screening Period.
- Open-Label - Placebo SC to Belimumab 200 mg SC: Par. received placebo administered SC once weekly through 51 weeks of the treatment period. Par. continued with the stable standard therapy they were receiving during the Screening Period. Par. who completed the Double-Blind phase with active SLE were assessed for eligibility to participate in a 6-month extension phase during which they received open label belimumab 200 mg SC weekly.
- Open-Label - Belimumab 200 SC to Belimumab 200 mg SC: Par. received belimumab 200 mg administered SC once weekly through 51 weeks of the treatment period. Par. continued with the stable standard therapy they were receiving during the Screening Period. Par. who completed the Double-Blind phase with active SLE were assessed for eligibility to participate in a 6-month extension phase during which they received open label belimumab 200 mg SC weekly
Period: Period 1
Arm/Group | Placebo SC | Belimumab 200 mg SC | Open-Label - Placebo SC to Belimumab 200 mg SC | Open-Label - Belimumab 200 SC to Belimumab 200 mg SC
Started | 280 | 556 | 0 | 0
Completed | 214 | 463 | 0 | 0
Not Completed | 66 | 93 | 0 | 0
Not completed — Protocol Violation | 3 | 4 | 0 | 0
Not completed — Physician Decision | 5 | 1 | 0 | 0
Not completed — Lack of Efficacy | 10 | 15 | 0 | 0
Not completed — Adverse Event | 25 | 40 | 0 | 0
Not completed — Withdrawal by Subject | 15 | 12 | 0 | 0
Not completed — Lost to Follow-up | 2 | 6 | 0 | 0
Not completed — Positive Pregnancy | 1 | 6 | 0 | 0
Not completed — Treatment Failure | 3 | 6 | 0 | 0
Not completed — Lack of Compliance | 2 | 1 | 0 | 0
Not completed — Unable to Visit Site | 0 | 2 | 0 | 0
Period: Period 2
Arm/Group | Placebo SC | Belimumab 200 mg SC | Open-Label - Placebo SC to Belimumab 200 mg SC | Open-Label - Belimumab 200 SC to Belimumab 200 mg SC
Started | 0 | 0 | 206 | 456
Completed | 0 | 0 | 191 | 434
Not Completed | 0 | 0 | 15 | 22
Not completed — Lack of Efficacy | 0 | 0 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 5 | 13
Not completed — Other | 0 | 0 | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Placebo SC: Par. received placebo administered SC, once weekly through 51 weeks of the treatment period. Par. continued with the stable standard therapy they were receiving during the Screening Period.
- Belimumab 200 mg SC: Par. received belimumab 200 mg administered SC once weekly through 51 weeks of the treatment period. Par. continued with the stable standard therapy they were receiving during the Screening Period.
- Total: Total of all reporting groups
Arm/Group | Placebo SC | Belimumab 200 mg SC | Total
Number analyzed (Participants) | 280 | 556 | 836
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.6 (12.61) | 38.1 (12.10) | 38.6 (12.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 268 | 521 | 789
  Male | 12 | 35 | 47
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian/European Heritage | 160 | 326 | 486
  Middle East/North African Heritage | 6 | 10 | 16
  Central Asian Heritage | 0 | 2 | 2
  East Asian Heritage | 15 | 29 | 44
  Japanese Heritage | 16 | 13 | 29
  South Asian Heritage | 0 | 2 | 2
  Southeast Asian Heritage | 32 | 73 | 105
  African American/African Heritage | 30 | 56 | 86
  American Indian or Alaska Native | 21 | 43 | 64
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Par. Achieving a SLE Responder Index (SRI) Response Rate at Week 52
Description: SRI response is defined as >=4 point reduction, from Baseline in safety of estrogen in lupus national assessment (SELENA) systemic lupus erythematosus disease activity index (SLEDAI) score, no worsening (increase of <0.30 points from Baseline) in physician's global assessment (PGA) and no new British Isles Lupus Assessment Group of SLE clinics (BILAG) A organ domain score or 2 new BILAG B organ domain scores compared with Baseline. Analysis was performed using a logistic regression model for the comparison between belimumab and placebo with covariates treatment group, Baseline SELENA SLEDAI score (<=9 vs. >=10), Baseline complement levels (low C3 and/or C4 vs. no low C3 or C4) and race (black vs. other).
Time Frame: Week 52
Population: Intention-To-Treat (ITT) Population: comprised of all par. who were randomized and treated with at least one dose of study treatment. Three par. did not have a Baseline PGA assessment; therefore, were not included.
Measure: Number; unit: Percentage of par.
Groups:
- Placebo SC: Par. received placebo administered SC once weekly through 51 weeks of the treatment period. Par. continued with the stable standard therapy they were receiving during the Screening Period.
Arm/Group | Placebo SC | Belimumab 200 mg SC
Number analyzed (Participants) | 279 | 554
Percentage of par. | 48.4 | 61.4
Statistical Analysis 1: Comparison: Placebo SC vs Belimumab 200 mg SC; Test type: Superiority or Other; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.25 to 2.25]

2. Secondary Outcome: Time to First Severe Flare (as Measured by the Modified SLE Flare Index)
Description: Time to first severe SLE flare is defined as the number of days from treatment start date until the participant met an event (event date - treatment start date +1). Analyses of severe SLE flare was performed on modified SELENA SLEDAI SLE flare index that excludes severe flares that were triggered only by an increase in SELENA SLEDAI score to >12 (since this may only represent a modest increase in disease activity). Only post-baseline severe flares were considered.
Time Frame: Baseline (Day 0, prior to dosing) to Week 52
Population: ITT population. Only those participants available at that particular timepoints were analyzed.
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo SC | Belimumab 200 mg SC
Number analyzed (Participants) | 51 | 59
Days | 118 [2 to 364] | 171 [5 to 358]
Statistical Analysis 1: Comparison: Placebo SC vs Belimumab 200 mg SC; Test type: Superiority or Other; p = 0.0004, Cox proportional hazards model; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.35 to 0.74]

3. Secondary Outcome: Percentage of Par. Whose Average Prednisone Dose Had Been Reduced by >=25% From Baseline to <=7.5 mg/Day During Weeks 40 Through 52 in Par. Receiving Greater Than 7.5 mg/Day at Baseline
Description: For the analysis of steroid use, all steroid dosages were converted to a prednisone equivalent in mg. The average daily prednisone dose was calculated taking into account all steroids taken intravenously, intramuscularly, SC, intradermally and orally for both SLE and non-SLE reasons. A responder was defined as having a prednisone reduction by >=25% from Baseline to <=7.5 mg/day during Weeks 40 through 52. At Baseline, the average daily prednisone dose was the sum of all prednisone doses over 7 consecutive days up to, but not including Day 0, divided by 7. For this analysis, the average prednisone dose was the total prednisone dose during weeks 40 through 52 divided by the number of days during Weeks 40 through 52. Analysis was performed using a logistic regression model with covariates treatment group, Baseline prednisone dose, Baseline SELENA SLEDAI score, (<=9 vs >=10), Baseline complement levels (low C3 and/or C4 vs. no low C3 or C4) and race (black vs. other).
Time Frame: Baseline (Day 0, prior to dosing), Weeks 40 through Week 52
Population: ITT population. Only par. with Baseline prednisone dose >7.5 mg/day were included.
Measure: Number; unit: Percentage of par.
Arm/Group | Placebo SC | Belimumab 200 mg SC
Number analyzed (Participants) | 168 | 335
Percentage of par. | 11.9 | 18.2
Statistical Analysis 1: Comparison: Placebo SC vs Belimumab 200 mg SC; Test type: Superiority or Other; p = 0.0732, Regression, Logistic; Odds Ratio (OR) = 1.65, 95% CI 2-sided [0.95 to 2.84]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-SAEs were collected from start of study drug administration to 51 weeks of treatment period/Exit visit for those par. who withdrew during double-blind treatment, plus another 6 months for open-label treatment period.
Description: SAEs and non-SAEs were collected in par. of ITT population, which comprised of par. who were randomized and treated with at least one dose of study treatment.
Arm/Group | Placebo SC | Belimumab 200 mg SC | Open-Label - Placebo SC to Belimumab 200 mg SC | Open-Label - Belimumab 200 SC to Belimumab 200 mg SC
All-Cause Mortality (participants affected / at risk) | 2/280 | 3/556 | 0/206 | 0/456
Serious Adverse Events (participants affected / at risk) | 44/280 | 60/556 | 14/206 | 25/456
Other Adverse Events (participants affected / at risk) | 218/280 | 403/556 | 42/206 | 78/456
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo SC (N=280) | Belimumab 200 mg SC (N=556) | Open-Label - Placebo SC to Belimumab 200 mg SC (N=206) | Open-Label - Belimumab 200 SC to Belimumab 200 mg SC (N=456)
Cellulitis (Infections and infestations) | 2 | 3 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 4 | 1 | 1
Pneumonia bacterial (Infections and infestations) | 2 | 3 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 3 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 2 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 2 | 0 | 1
Amoebic dysentery (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Corynebacterium sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
External ear cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 2 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Osteomyelitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 1
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 1 | 0
Tuberculosis of central nervous system (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 4 | 0 | 0
Lupus nephritis (Renal and urinary disorders) | 1 | 2 | 0 | 0
Nephritis (Renal and urinary disorders) | 1 | 2 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 2 | 0 | 1 | 0
Nephritic syndrome (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0
Neuropsychiatric lupus (Nervous system disorders) | 0 | 2 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0
Intracranial venous sinus thrombosis (Nervous system disorders) | 0 | 1 | 0 | 0
Lupus encephalitis (Nervous system disorders) | 1 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
SLE arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 3 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 1 | 2
Lupus vasculitis (Vascular disorders) | 2 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lipoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Exfoliation syndrome (Eye disorders) | 0 | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 1 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lupus pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Central nervous system lupus (Nervous system disorders) | 0 | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 2 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 1 | 0
Mycobacterial infection (Infections and infestations) | 0 | 0 | 1 | 0
Paraspinal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1
Polycystic ovaries (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo SC (N=280) | Belimumab 200 mg SC (N=556) | Open-Label - Placebo SC to Belimumab 200 mg SC (N=206) | Open-Label - Belimumab 200 SC to Belimumab 200 mg SC (N=456)
Viral upper respiratory tract infection (Infections and infestations) | 24 | 48 | 9 | 17
Nasopharyngitis (Infections and infestations) | 22 | 38 | 9 | 7
Urinary tract infection bacterial (Infections and infestations) | 18 | 41 | 2 | 14
Upper respiratory tract infection bacterial (Infections and infestations) | 14 | 30 | 3 | 9
Nausea (Gastrointestinal disorders) | 22 | 38 | 1 | 5
Diarrhoea (Gastrointestinal disorders) | 14 | 27 | 3 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 28 | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 31 | 6 | 11
Headache (Nervous system disorders) | 25 | 57 | 4 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 22 | 1 | 8
Insomnia (Psychiatric disorders) | 20 | 18 | 0 | 1
Hypertension (Vascular disorders) | 14 | 25 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.